CLINICAL TRIAL: NCT05466292
Title: Evaluation of a Clinical Ethics Committee (CEC) Implementation Process in an Oncological Research Hospital. A Process Evaluation Study Using Normalization Process Theory
Brief Title: Evaluating a Clinical Ethics Committee (CEC) Implementation Process
Acronym: Val_CEC
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1085/2021/OSS/IRCCSRE
Record Dates: First submitted 2022-07-14; First posted 2022-07-20 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Service Evaluation
Keywords: Ethics Committees, Clinical; Evaluation Studies as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthcare Professionals (HPs) employed at the Local Health Authority of Reggio Emilia,: HPs will be included if they are employed at the Health Care Authority of Reggio Emilia. They will receive a closed-ended questions survey.
  Interventions: Other: Survey1
- Local Health Authority's Managers/Wards Heads: Managers/Heads who formally supported and promoted the intervention or have been contacted during the dissemination process will be interviewed by semi-structured interview.
  Interventions: Other: semi-structured interview_1
- Clinical Ethics Committee (CEC)'s members: CEC's members will be interviewed by semi-structured interview.
  Interventions: Other: semi-structured interview_2
- Healthcare Professionals who submitted an ethics consultation request: Healthcare Professionals who submitted an ethics consultation request will be interviewed by semi-structured interview.
  Interventions: Other: semi-structured interview_3
- Healthcare Professionals who attended the training provided by the Clinical Ethics Committee: Healthcare Professionals who attended at least one of the five training courses on ethics consultation provided by the Clinical Ethics Committee. They will receive a survey of 20 multiple-choice questions and supplemented by free-text questions.
  Interventions: Other: survey_2

INTERVENTIONS:
Other: Survey1 — Closed-ended survey on the level of knowledge, use, and dissemination of the CEC.
  Groups: Healthcare Professionals (HPs) employed at the Local Health Authority of Reggio Emilia,
Other: semi-structured interview_1 — the semi-structured interview concerns participants'motivations/expectations for implementing CEC, personal attitude towards the service, experience with CEC in terms of facilitators, problems, and critical evaluation on the service delivered
  Groups: Local Health Authority's Managers/Wards Heads
Other: semi-structured interview_2 — semi-structured interview concerns participants motivations and expectations to be a member of the CEC, personal attitude towards the service, experience with CEC in terms of facilitators, problems, and critical evaluation on the service delivered.
  Groups: Clinical Ethics Committee (CEC)'s members
Other: semi-structured interview_3 — semi-structured interview concerns participants' experiences with the ethics consultation service provide by the Clinical Ethics Committee
  Groups: Healthcare Professionals who submitted an ethics consultation request
Other: survey_2 — survey of 20 multiple-choice questions and supplemented by free-text questions.
  Groups: Healthcare Professionals who attended the training provided by the Clinical Ethics Committee

SUMMARY:
This is a Mixed-method study with retrospective quantitative assessment and prospective qualitative evaluation focused on the development and implementation of a multidisciplinary Clinical Ethics Committee (CEC), 16 months from its implementation.

A CEC is a multi-professionals service that aims to support healthcare professionals (HPs) and healthcare organizations in dealing with ethical issues of clinical practice, providing also ethics consultations (EC) for complex clinical cases, characterized by conflicting ethical perspectives.

In 2020, a CEC was established in an Oncology Research Hospital in the North of Italy. It was developed and implemented according to the Medical Research Council (MRC) framework for developing and evaluating complex interventions.

The purpose of this study is to evaluate the CEC's development and implementation process, after 16 months it entered into force.

Study's hypothesis: the investigators expect to identify the relevant components that contribute to the CEC's successful implementation and integration into everyday practice. Findings would also identify required modifications to improve the service and develop practical strategies for enabling and sustaining the CEC delivery in clinical settings.

DETAILED DESCRIPTION:
The investigators will combine quantitative and qualitative methods to collect data on crucial process variables, from sites or participants purposively selected along such elements expected to influence the intervention's functioning.

The study consists of a quantitative and qualitative evaluation.

Quantitative evaluation. It aims to assess the CEC's activities performed within 16 months since its implementation and the spread, use, and knowledge of the service by all the HPs employed at the Local Health Authority of Reggio Emilia. These data will be used to examine the quantity of intervention implemented, and whether and how the intended audience came into contact with the intervention.

Data related to the amount of CEC activities will be collected by the internal database developed by the CEC Secretariat. Moreover, to collect data on the level of knowledge, use, and dissemination of the CEC, a closed-ended questions survey will be disseminated among all the HPs employed at the Oncology Research Hospital. Quantitative data will be analyzed using descriptive techniques.

Qualitative Evaluation. The qualitative evaluation aims to investigate mechanisms of impact and contextual factors among several groups of stakeholders, differently involved in designing, promoting, delivering, and benefitting the CEC. The Normalization Process Theory (NPT) will be applied to determine if, and in what ways, the CEC can be successfully 'normalized' into clinical practice. NPT is a theory aimed at identifying, characterizing, and explaining the empirically identifiable mechanism that motivates and shapes the implementation process of a complex intervention by four conceptual tools (coherence, cognitive participation, collective action, and reflexive monitoring). The NPT will inform the data collection tools of the qualitative part and will be used as a framework for data analysis.

Semi-structured interviews will be performed with different groups of stakeholders. The interviews' topics concern the 4 concepts of the NPT. A specific interview track will be developed for each interviewed group. Moreover, a second online survey will be sent to HPs who have attended at least 1 of the 5 editions of the ethics training promoted by the CEC. The survey will consist of 20 multiple-choice questions, also based on the constructs of the NPT, and will be supplemented by free-text questions aimed at assessing: the acceptability of the CEC within the local context and understanding additional needs and expectations about the service. Qualitative data will be thematically analyzed. After an initial inductive analysis of the qualitative data, the NPT concepts will be applied to the emerging themes to confirm or refine the results.

Ethical Considerations. Eligible subjects may only be included in the study after providing written informed consent. No study procedure can be performed before it has been provided.

ELIGIBILITY:
Inclusion Criteria:

* being a healthcare professionals (HPs) (physicians, therapists, nurses, social workers, healthcare researcher, pharmacist..)
* being an HPs employed at the Health Care Authority of Reggio Emilia;

Participants will be included in the qualitative evaluation if they:

* are working as a Head of Departments / local Manager at the Local health Authority of Reggio Emilia, and have been contacted by the CEC's President during the dissemination process;
* have been a member of the CEC in the last 16 months;
* submitted at least 1 ethics consultation request;
* participated to at least 1 of the 5 training courses on ethics consultation promoted by the CEC

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from Healthcare professionals employed at the local Health Authority of Reggio Emilia.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Process Evaluation by a quantitative, closed-ended questions surveys and semi-structured interviews with different groups of the Clinical Ethics Committee (CEC)'s stakeholders. | 16 months from the service implementation
  The evaluation of the development and implementation process of the CEC will be assessed quantitatively by assessing the activity of the CEC and its diffusions, knowledge and utilization among HPs, while qualitatively, by collecting the opinions and perspectives on it from users and provider healthcare professionals, in terms of perceived barriers/facilitators, expectations and needs towards the service.

SECONDARY OUTCOMES:
7 - issues CEC Survey | 16 months from service implementation
  It is a closed-ended survey aiming to collect information on the level of knowledge, use, and dissemination of the CEC among all the HPs employed at the Local Health Authority of Reggio Emilia.
  It is composed by 3 sections: section A asking participant's general information; section B asking participant's previous experience in ethical complex situation; section C asking patient's evaluation of the service in terms of: diffusion, knowledge, access, personal attitude, further suggestions.
  Answer are organized into Yes/No or free space.
semi-structured one-to-one interview | 16 months from service implementation
  semi-structured one-to-one interviews to explore the opinions and perspectives on the CEC, in terms of barriers/facilitators, expectations and needs, from the perspectives of Local Health Authority's Managers/Wards Heads who have been involved in the design and delivery of the service.
semi-structured one-to-one interview | 16 months from service implementation
  semi-structured one-to-one interviews with CEC's members' concerns their motivations and expectations to be a member of the CEC, personal attitude toward the service, experience with CEC in terms of facilitators, problems, and critical evaluation of the service delivered.
semi-structured interview with HPs who required ethics consultation | 16 months from service implementation
  semi-structured interview concerns participants' experiences with the ethics consultation service provide by the Clinical Ethics Committee
Normalisation MeAsure Development questionnaire (NoMAD) | 16 months from service implementation
  The NoMAD survey is a set of 20 survey items for assessing implementation processes from the perspective of professionals directly involved in the work of implementing complex interventions in healthcare. This version comprises 20 multiple-choice questions, supplemented by 4 open questions. Answers are organized into a range of 5 options : 1. I do not agree, 2. I partially not agree, 3. I do not agree or disagree, 4. I partially agree, 5. I totally agree. Higher scores mean better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Perin, MA, Principal Investigator — Azienda USL - IRCCS di Reggio Emilia
Locations (1):
- Azienda USL-IRCCS di Reggio Emilia, Reggio Emilia, Italia, Italy

IPD SHARING:
Plan to Share IPD: No
All the IPD will be anonimyzed. PErsonal data will be collected in an aggregate way to be shared within research publications.

REFERENCES:
- [Derived] Perin M, Magelssen M, Ghirotto L, De Panfilis L. Evaluating a clinical ethics committee (CEC) implementation process in an oncological research hospital: protocol for a process evaluation study using normalisation process theory (EvaCEC). BMJ Open. 2023 Mar 9;13(3):e067335. doi: 10.1136/bmjopen-2022-067335. PMID 36894200

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT05466292/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT05466292/ICF_002.pdf